CLINICAL TRIAL: NCT05855980
Title: Toe Amputations in Patients With Diabetes - the Effect of Leaving a Wound Open or Closing on Healing and Ambulation After Surgery.
Brief Title: Toe Amputations in Patients With Diabetes
Acronym: PANDORAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Miska Vuorlaakso, Principal Investigator, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R22101
Record Dates: First submitted 2023-04-05; First posted 2023-05-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Foot; Infections; Amputation
Keywords: Diabetic foot; Infection; Amputation
MeSH Terms: conditions — Diabetic Foot; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed wound (Active Comparator): Wound is closer immediately after amputation (instead healing secondarily)
  Interventions: Procedure: Wound closure
- Open wound (No Intervention): Wound is left to heal secondarily

INTERVENTIONS:
Procedure: Wound closure — Wound is closed or left open to heal secondarily after amputation.
  Arms: Closed wound

SUMMARY:
This study is a randomized controlled trial (RCT) to evaluate outcome after toe amputation due to diabetic foot infection. Aim of this RCT is to evaluate wound healing and functional outcome based, whether wound is closed or left open. As a part of this study, emerging technology of thermal imaging is evaluated as a possible tool to predict complication after amputation.

DETAILED DESCRIPTION:
Patients with diabetes undergoing toe amputation due to infection, are recruited for this study. Based on randomization, wound is either closed or left open during the amputation procedure. If primary closure is not possible (e.g. deep abscess) and patient is randomized to closed group, delayed closure is performed when feasible. Patients are followed up in outpatient clinic 3 month after amputation. Primary outcome is wound healing that is evaluated during follow ups in the outpatient clinic. Functional outcome is evaluated with PROM questionnaires preoperatively and during the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Toe amputation due to diabetic foot infection

Exclusion Criteria:

* Deep foot infection
* Sepsis
* No clinical infection (amputation due to trauma, deformity or uninfected necrosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Wound healed | 3 months
  Percentage of patients with completely healed (no dehiscence, necrosis etc.) wound in 3 month control visit

SECONDARY OUTCOMES:
Complications | 3 months
  Percentage of patients experiencing complication during 3 month follow-up
Functional outcome: 15D | 3 months
  15D quality of life questionnaire 3 months after amputation and change compared to preoperative 15D score.
  15D is 15 dimensional questionnaire that provides score between 0 and 1 representing health related quality of life (HRQOL). Higher value represents better HRQOL.
Functional outcome: TESS | 3 months
  Toronto extremity salvage score (TESS) questionnaire 3 months after amputation and change compared to preoperative TESS score.
  TESS is contains 30 questions (rated 1-5) measuring activity limitations. TESS result is a percentage of the maximum score, 100 representing normal activity.
Functional outcome: FHSQ | 3 months
  Foot health status questionnaire (FHSQ) 3 months after amputation and change compared to preoperative FHSQ score.
  FHSQ consists of 19 questions that ultimately provide score 0-100 higher value representing better foot health status.

CONTACTS AND LOCATIONS:
Overall Officials: Miska Vuorlaakso, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland